CLINICAL TRIAL: NCT02607735
Title: A Phase 3, Global, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir/GS-9857 Fixed-Dose Combination for 12 Weeks in Direct-Acting Antiviral-Experienced Subjects With Chronic HCV Infection
Brief Title: Safety and Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir in Adults With Chronic HCV Infection Who Have Previously Received Treatment With Direct-Acting Antiviral Therapy
Acronym: POLARIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-367-1171; 2015-003455-21 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SOF/VEL/VOX (Primary Study) (Experimental): SOF/VEL/VOX for 12 weeks
  Interventions: Drug: SOF/VEL/VOX
- Placebo (Primary Study) (Experimental): Placebo to match SOF/VEL/VOX for 12 weeks
  Interventions: Drug: Placebo
- SOF/VEL/VOX (Deferred Treatment Substudy) (Experimental): SOF/VEL/VOX for 12 weeks for eligible participants initially randomized to receive placebo
  Interventions: Drug: SOF/VEL/VOX

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg fixed dose-combination (FDC) tablet administered orally once daily with food
  Other Names: Vosevi®; GS-7977/GS-5816/GS-9857
  Arms: SOF/VEL/VOX (Deferred Treatment Substudy); SOF/VEL/VOX (Primary Study)
Drug: Placebo — Tablet administered orally once daily with food
  Arms: Placebo (Primary Study)

SUMMARY:
The primary objectives of this study are to evaluate the safety and efficacy of treatment with sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) in adults with chronic hepatitis C virus (HCV) infection who have previously received treatment with direct-acting antiviral therapy.

Participants randomized to placebo may be eligible for deferred treatment with active SOF/VEL/VOX.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic HCV infection (≥ 6 months)
* Treatment experienced with a direct acting antiviral medication for HCV
* Use of protocol specified methods of contraception

Key Exclusion Criteria:

* Current or prior history of clinically significant illness that may interfere with participation in the study
* Screening ECG with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at screening
* Pregnant or nursing female
* Chronic liver disease not caused by HCV
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (86):
- United States (43):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Pasadena, California
  - Rialto, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Catonsville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - New York, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (6):
  - Camperdown, New South Wales
  - Darlinghurst, New South Wales
  - Herston, Queensland
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Melbourne, Victoria
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brampton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (18):
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Rennes
  - Rouen
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (6):
  - Berlin
  - Bonn
  - Cologne
  - Frankfurt am Main
  - Hamburg
  - Hanover
- New Zealand (2):
  - Christchurch
  - Grafton
- San Juan, Puerto Rico
- United Kingdom (4):
  - London
  - Manchester
  - Nottingham
  - Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Background] Bourlière M, Gordon SC, Ramji A, Ravendhran N, Tran TT, Hyland RH, et al. Sofosbuvir/Velpatasvir/Voxilaprevir for 12 Weeks as a Salvage Regimen in NS5A Inhibitor-Experienced Patients with Genotype 1-6 Infection: The Phase 3 POLARIS-1 Study [Abstract 194]. J Hepatology 2016;63 (1S):102A.
- [Background] Younossi ZM, Stepanova M, Gordon S, Zeuzem S, Mann MP, Jacobson I, Bourliere M, Cooper C, Flamm S, Reddy KR, Kowdley K, Younossi I, Hunt S. Patient-Reported Outcomes Following Treatment of Chronic Hepatitis C Virus Infection With Sofosbuvir and Velpatasvir, With or Without Voxilaprevir. Clin Gastroenterol Hepatol. 2018 Apr;16(4):567-574.e6. doi: 10.1016/j.cgh.2017.11.023. Epub 2017 Nov 16. PMID 29155352
- [Background] Bourliere M, Gordon SC, Schiff ER, Tran TT, Ravendhran N, Landis CS, Hyland RH, Stamm LM, Zhang J, Dvory-Sobol H, Subramanian GM, Brainard DM, McHutchison JG, Serfaty L, Thompson AJ, Sepe TE, Curry MP, Reddy KR, Manns MP. Deferred treatment with sofosbuvir-velpatasvir-voxilaprevir for patients with chronic hepatitis C virus who were previously treated with an NS5A inhibitor: an open-label substudy of POLARIS-1. Lancet Gastroenterol Hepatol. 2018 Aug;3(8):559-565. doi: 10.1016/S2468-1253(18)30118-3. Epub 2018 May 31. PMID 29859740
- [Result] Bourliere M, Gordon SC, Flamm SL, Cooper CL, Ramji A, Tong M, Ravendhran N, Vierling JM, Tran TT, Pianko S, Bansal MB, de Ledinghen V, Hyland RH, Stamm LM, Dvory-Sobol H, Svarovskaia E, Zhang J, Huang KC, Subramanian GM, Brainard DM, McHutchison JG, Verna EC, Buggisch P, Landis CS, Younes ZH, Curry MP, Strasser SI, Schiff ER, Reddy KR, Manns MP, Kowdley KV, Zeuzem S; POLARIS-1 and POLARIS-4 Investigators. Sofosbuvir, Velpatasvir, and Voxilaprevir for Previously Treated HCV Infection. N Engl J Med. 2017 Jun 1;376(22):2134-2146. doi: 10.1056/NEJMoa1613512. PMID 28564569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia Pacific. The first participant was screened on 11 November 2015. The last study visit occurred on 21 June 2017.
Pre-assignment Details: 520 participants were screened.
Groups:
- SOF/VEL/VOX (Primary Study): Sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) (400/100/100 mg) fixed-dose combination (FDC) tablet orally once daily with food for 12 weeks
- Placebo (Primary Study): Placebo tablet orally once daily with food for 12 weeks
- SOF/VEL/VOX (Deferred Treatment Substudy): Participants who completed placebo treatment were eligible to enroll in to the open-label Deferred Treatment Substudy to receive SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 12 weeks.
Period: Primary Study
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study) | SOF/VEL/VOX (Deferred Treatment Substudy)
Started | 264 | 152 | 0
Completed | 257 | 152 | 0
Not Completed | 7 | 0 | 0
Not completed — Randomized but Never Treated | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Withdrew Consent | 2 | 0 | 0
Period: Deferred Treatment Substudy
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study) | SOF/VEL/VOX (Deferred Treatment Substudy)
Started | 0 | 0 | 147
Completed | 0 | 0 | 142
Not Completed | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Withdrew Consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug
Groups:
- SOF/VEL/VOX (Primary Study): SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study) | Total
Number analyzed (Participants) | 263 | 152 | 415
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8.5) | 59 (8.0) | 58 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 31 | 94
  Male | 200 | 121 | 321
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 211 | 124 | 335
  Black or African American | 38 | 22 | 60
  Asian | 8 | 6 | 14
  Native Hawaiian or Pacific Islander | 3 | 0 | 3
  Not Disclosed | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 247 | 142 | 389
  Not Disclosed | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 135 | 101 | 236
  Australia | 15 | 11 | 26
  Canada | 28 | 14 | 42
  France | 56 | 16 | 72
  Germany | 16 | 7 | 23
  New Zealand | 5 | 2 | 7
  United Kingdom | 8 | 1 | 9
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene
  Participants
    CC | 47 | 27 | 74
    CT | 165 | 93 | 258
    TT | 51 | 32 | 83
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.68) | 6.3 (0.63) | 6.3 (0.66)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 73 | 36 | 109
  ≥ 800,000 IU/mL | 190 | 116 | 306

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12) (Primary Study)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Participants in the Full Analysis Set (all randomized/enrolled participants who took at least 1 dose of study drug) in the SOF/VEL/VOX group were analyzed. This outcome measure was not assessed for participants in the Placebo group because they did not have a Posttreatment Week 12 visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Primary Study)
Number analyzed (Participants) | 263
percentage of participants | 96.2 [93.1 to 98.8]
Statistical Analysis 1: Comparison: SOF/VEL/VOX (Primary Study); Test type: Superiority — The SVR12 rate for the SOF/VEL/VOX group was compared to the performance goal of 85% using a 2-sided exact 1-sample binomial test at the 0.05 significance level; p < 0.001, 2-sided exact 1-sample binomial test

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event (Primary Study)
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study)
Number analyzed (Participants) | 263 | 152
percentage of participants | 0.4 | 2.0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4) (Primary Study)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study)
Number analyzed (Participants) | 263 | 152
percentage of participants | 97.7 [95.1 to 99.2] | 0 [0.0 to 2.4]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment (Primary Study)
Time Frame: Weeks 1, 2, 4, 8 and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study)
Number analyzed (Participants) | 263 | 152
percentage of participants
  Week 1 | 15.6 [11.4 to 20.5] | 0 [0.0 to 2.4]
  Week 2: number analyzed (Participants) | 263 | 150
  Week 2 | 56.7 [50.4 to 62.7] | 0 [0.0 to 2.4]
  Week 4: number analyzed (Participants) | 262 | 150
  Week 4 | 92.7 [88.9 to 95.6] | 0 [0.0 to 2.4]
  Week 8: number analyzed (Participants) | 262 | 150
  Week 8 | 100.0 [98.6 to 100.0] | 0 [0.0 to 2.4]
  Week 12: number analyzed (Participants) | 261 | 149
  Week 12 | 99.6 [97.9 to 100.0] | 0 [0.0 to 2.4]

5. Secondary Outcome: Change From Baseline in HCV RNA (Primary Study)
Time Frame: Baseline; Weeks 1, 2, 4, 8 and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study)
Number analyzed (Participants) | 262 | 150
log10 IU/mL
  Week 1: number analyzed (Participants) | 258 | 150
  Week 1 | -4.20 (0.733) | 0.02 (0.300)
  Week 2: number analyzed (Participants) | 261 | 148
  Week 2 | -4.81 (0.704) | 0.02 (0.322)
  Week 4: number analyzed (Participants) | 261 | 150
  Week 4 | -5.07 (0.677) | -0.01 (0.441)
  Week 8: number analyzed (Participants) | 262 | 149
  Week 8 | -5.11 (0.678) | 0.05 (0.434)
  Week 12: number analyzed (Participants) | 261 | 138
  Week 12 | -5.10 (0.690) | 0.03 (0.430)

6. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24) (Primary Study)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set in the SOF/VEL/VOX group were analyzed. This outcome measure was not assessed for participants in the Placebo group because they did not have a Posttreatment Week 24 visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Primary Study)
Number analyzed (Participants) | 263
percentage of participants | 96.2 [93.1 to 98.2]

7. Secondary Outcome: Percentage of Participants With Virologic Failure (Primary Study)
Description: Virologic failure is defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA LLOQ while on treatment), or
    * Rebound (confirmed 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Primary Study)
Number analyzed (Participants) | 263
percentage of participants | 2.7

8. Secondary Outcome: Percentage of Participants With SVR at 4, 12, and 24 Weeks After Discontinuation of Therapy (Deferred Treatment Substudy)
Description: SVR4, SVR12 and SVR24 was defined as HCV RNA < LLOQ at 4, 12 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4, 12, and 24 (Deferred Treatment Substudy)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL/VOX (Deferred Treatment Substudy): SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 12 weeks
Arm/Group | SOF/VEL/VOX (Deferred Treatment Substudy)
Number analyzed (Participants) | 147
percentage of participants
  SVR4 | 98.6 [95.2 to 99.8]
  SVR12 | 97.3 [93.2 to 99.3]
  SVR24 | 97.3 [93.2 to 99.3]

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment (Deferred Treatment Substudy)
Time Frame: Weeks 1, 2, 4, 8 and 12 (Deferred Treatment Substudy)
Population: Full Analysis Set from the Deferred Treatment Sub study: all enrolled participants who took at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Deferred Treatment Substudy)
Number analyzed (Participants) | 147
percentage of participants
  Week 1 | 14.3 [9.1 to 21.0]
  Week 2 | 62.6 [54.2 to 70.4]
  Week 4 | 93.2 [87.8 to 96.7]
  Week 8 | 100.0 [97.5 to 100.0]
  Week 12 | 100.0 [97.5 to 100.0]

10. Secondary Outcome: Change From Baseline in HCV RNA (Deferred Treatment Substudy)
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12 (Deferred Treatment Substudy)
Population: Participants with available data in the Full Analysis Set of the Deferred Treatment Substudy were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX (Deferred Treatment Substudy)
Number analyzed (Participants) | 147
log10 IU/mL
  Week 1: number analyzed (Participants) | 139
  Week 1 | -4.30 (0.626)
  Week 2: number analyzed (Participants) | 145
  Week 2 | -4.93 (0.602)
  Week 4 | -5.16 (0.512)
  Week 8 | -5.20 (0.532)
  Week 12 | -5.20 (0.532)

11. Secondary Outcome: Percentage of Participants With Virologic Failure (Deferred Treatment Substudy)
Description: as for outcome 7
Time Frame: Up to Posttreatment Week 24 (Deferred Treatment Substudy)
Population: Full Analysis Set in the Deferred Treatment Substudy
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX (Deferred Treatment Substudy)
Number analyzed (Participants) | 147
percentage of participants | 2.7

ADVERSE EVENTS:
Time Frame: Primary Study: Up to 12 Weeks + 30 days; Deferred Treatment Substudy: Up to 12 Weeks + 30 days
Description: Safety Analysis Set: all participants who received at least 1 dose of study drug
Groups:
- SOF/VEL/VOX (Deferred Treatment Substudy): Participants who completed placebo treatment were eligible for open-label Deferred Treatment Substudy.
  SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 12 weeks
Arm/Group | SOF/VEL/VOX (Primary Study) | Placebo (Primary Study) | SOF/VEL/VOX (Deferred Treatment Substudy)
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/152 | 0/147
Serious Adverse Events (participants affected / at risk) | 5/263 | 7/152 | 6/147
Other Adverse Events (participants affected / at risk) | 147/263 | 80/152 | 87/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX (Primary Study) (N=263) | Placebo (Primary Study) (N=152) | SOF/VEL/VOX (Deferred Treatment Substudy) (N=147)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arteritis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX (Primary Study) (N=263) | Placebo (Primary Study) (N=152) | SOF/VEL/VOX (Deferred Treatment Substudy) (N=147)
Diarrhoea (Gastrointestinal disorders) | 48 | 19 | 28
Nausea (Gastrointestinal disorders) | 37 | 12 | 21
Asthenia (General disorders) | 20 | 9 | 3
Fatigue (General disorders) | 56 | 30 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 7
Dizziness (Nervous system disorders) | 11 | 14 | 7
Headache (Nervous system disorders) | 66 | 26 | 29
Insomnia (Psychiatric disorders) | 19 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years